CLINICAL TRIAL: NCT03956303
Title: Comparison of the Efficacy of 3 Different Density Levobupivacaine Solutions + Fentanyl Applied Intrathecally for Spinal Anesthesia in Caesarean Delivery.
Brief Title: Comparison of 3 Different Density Levobupivacaine Solutions + Fentanyl for Spinal Anaesthesia for Caesarean Delivery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ozlem Sagir, MD, Associated Professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: osagir2
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia
Keywords: Anesthesia, Spinal; Cesarean Section; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Plain Levobupivacaine (Chirocaine (% 0.5) (Active Comparator): Levobupivacaine 8 mg (Chirocaine (% 0.5)) + 20 mcg fentanyl Chirocaine Plain
  Interventions: Drug: Chirocaine %0.5
- Levobupivacaine (Chirocaine % 0,75) + dextrose 40 (Active Comparator): Levobupivacaine 8 mg (Chirocaine % 0,75) + 20 mcg fentanyl + dextrose 40 Chirocaine Heavy 40
  Interventions: Drug: Chirocaine Heavy 40
- Levobupivacaine (Chirocaine % 0,75) + dextrose 60 (Active Comparator): Levobupivacaine 8 mg (Chirocaine % 0,75) + 20 mcg fentanyl + dextrose 60 Chirocaine Heavy 60
  Interventions: Drug: Chirocaine Heavy 60
- Levobupivacaine (Chirocaine % 0,75) + dextrose 80 (Active Comparator): Levobupivacaine 8 mg (Chirocaine % 0,75) + 20 mcg fentanyl + dextrose 80 Chirocaine Heavy 80
  Interventions: Drug: Chirocaine Heavy 80

INTERVENTIONS:
Drug: Chirocaine %0.5 — Levobupivacaine 8 mg Chirocaine (% 0.5) +20 mcg fentanyl
  Other Names: Plain levobupivacaine; Group 1
  Arms: Plain Levobupivacaine (Chirocaine (% 0.5)
Drug: Chirocaine Heavy 40 — Chirocaine (%0.75) + Dextrose 40 mg+20 mcg fentanyl
  Other Names: levobupivacaine heavy 40; Group 2
  Arms: Levobupivacaine (Chirocaine % 0,75) + dextrose 40
Drug: Chirocaine Heavy 60 — Chirocaine (%0.75) + Dextrose 60 mg+20 mcg fentanyl
  Other Names: levobupivacaine heavy 60; Group 3
  Arms: Levobupivacaine (Chirocaine % 0,75) + dextrose 60
Drug: Chirocaine Heavy 80 — Chirocaine (%0.75) + Dextrose 80 mg+20 mcg fentanyl
  Other Names: levobupivacaine heavy 80; Group 4
  Arms: Levobupivacaine (Chirocaine % 0,75) + dextrose 80

SUMMARY:
The investigator's aim is to compare the efficacy of 3 levobupivacaine solutions with different density on spinal anesthesia for caesarean delivery.

DETAILED DESCRIPTION:
Patients scheduled for elective caesarean delivery were separated into 4 groups. Spinal anesthesia was performed with one of the following regimens.

Group 1: Levobupivacaine 8 mg + 20 mcg Fentanyl Group 2: Levobupivacaine 8 mg + 20 mcg Fentanyl + 40 mg Dextrose Group 3: Levobupivacaine 8 mg + 20 mcg Fentanyl + 60 mg Dextrose Group 4: Levobupivacaine 8 mg + 20 mcg Fentanyl + 80 mg Dextrose After anesthesia induction motor block was evaluated via bromage scale and sensory block via pinprick test every 3 minutes for the first 15 minutes, and every 5 minutes up to 60 minutes. Maximum sensory block level, time to reach maximum block level, time needed to achieve T10 sensory level were recorded.

Baby delivery time, and operation duration were also recorded. Time to two segment regression of maximum sensory block, motor block recovery time and time to S2 regression of sensory block will be recorded.

Hemodynamic data, nausea vomiting, were also recorded throughout surgery at the same evaluation periods and postoperative period.

The surgeon will also evaluate the abdominal relaxation surgical block quality as good, medium and poor.

The patient will evaluate spinal block analgesia quality as good, medium or poor.

Pain scores are going to be evaluated by VAS at the beginning, uterine incision and during abdominal closure. Time for first analgesic requirement and postoperative pain is also going to be evaluated by VAS.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Pregnancy at Term
* Scheduled for elective caesarean delivery

Exclusion Criteria:

* contraindication for spinal anesthesia
* drug allergy
* pregnancy related disorders (hypertension, placenta previa, fetal problems)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change of time to reach T10 sensory spinal block level at intraoperative period by pinprick test | Every 3 minutes for 15 minutes and every 5 minutes afterwards up to 60 minutes after induction of spinal anesthesia.In these evaluation periods, the sensory block will be recorded when the T10 is detected.
  time to reach T10 sensory block by pinprick test
Spinal Block Quality by questioning | At the end of surgery
  the intensity of spinal block will be evaluated via questioning the surgeon and the patient. the surgeon will grade the abdominal relaxivity as good, medium or poor The patient will evaluate spinal block analgesia quality as good, medium or poor.
Change the sensory block level at intraoperative period by pinprick test | Every 3 minutes for 15 minutes and every 5 minutes afterwards up to 60 minutes after induction of spinal anesthesia. The highest measured level by pinprick test be recorded
  the level of maximum sensory block by pinprick test
time to reach maximum level of sensory block at intraoperative period by pinprick test | Every 3 minutes for 15 minutes and every 5 minutes afterwards up to 60 minutes after induction of spinal anesthesia. the time to reach the highest measured by pinprick test will be recorded.
  time to reach maximum level of sensory block by pinprick test
Change over time at the level of sensory block at intraoperative period by pinprick test | Every 3 minutes for 15 minutes and every 5 minutes afterwards up to 60 minutes after induction of spinal anesthesia. The time to two segment regression of maximum sensory block by pinprick test will be recorded.
  time to two segment regression of maximum sensory block by pinprick test
Change in motor block level from PACU to discharge | every 15 minutes until end of surgery and 30 minutes postoperatively up to 2 hours by Bromage Scale
  motor block recovery time by bromage scale
Change to regression of sensory block by pinprick test | In the postoperative period, changes in sensory block level will be recorded at 30 min intervals up to 2 hours
  time to S2 regression of sensory block by pinprick test

SECONDARY OUTCOMES:
Haemodynamic evaluation by mmHg for systolic , diastolic and mean arterial blood pressure | Every 3 minutes for 15 minutes and every 5 minutes afterwards up to 60 minutes after induction of spinal anesthesia. every 30 minutes up to 2 hours
  measurement of systolic , diastolic and mean arterial blood pressure
Number of participants with postoperative complications ( head ache, back pain, numbness of lower extremity )by phone | on postoperative day 3 by phone.
  postoperative complications ( head ache, back pain, numbness of lower extremity )by phone
evaluation of umbilical vein blood gas analysis | immediately after fetus delivery
  umbilical vein blood sample will be obtained immediately after delivery of the fetus and will a blood gas analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Sagir, Assist. Prof, Study Director — Balikesir University School of Medicine Department of Anesthesia and Reanimation